CLINICAL TRIAL: NCT01524770
Title: Comparative Pharmacokinetics of Dulaglutide After Administration Via an Auto-injector and a Manual Syringe in Healthy Subjects
Brief Title: A Study to Compare the Effect of Giving Dulaglutide Using an Auto-injector Versus a Manual Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14142; H9X-MC-GBDT (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual syringe (Active Comparator): Dulaglutide: Single dose of 1.5 milligrams (mg) dulaglutide administered subcutaneously (SC) by manual syringe in one of two study periods separated by a 28-day minimum washout period.
  Interventions: Biological: Dulaglutide
- Auto-injector (Experimental): Dulaglutide: Single dose of 1.5 milligrams (mg) dulaglutide administered subcutaneously (SC) by auto-injector in one of two study periods separated by a minimum 28-day washout period
  Interventions: Biological: Dulaglutide

INTERVENTIONS:
Biological: Dulaglutide — Administered by subcutaneous (SC) injection
  Other Names: LY2189265

SUMMARY:
The study involves 2 injections of 1.5 milligrams (mg) dulaglutide, 1 given by a pre-filled manual syringe, the other given by an auto-injector. Injections will be separated by a minimum 28-day washout period. The study will evaluate if the levels of drug in the blood are similar when given by each method. Participation in the study is likely to take approximately 7 weeks, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Male participants with female partners of child-bearing potential or partners who are pregnant or breastfeeding agree to use a reliable method of contraception from the time of the first dose until 3 months after the last dose of investigational product, as determined by the investigator
* The method may be one of the following:

  * condom with spermicidal agent
  * male participant sterilization
  * true abstinence (which is in line with the participant's usual lifestyle choice; withdrawal or calendar methods are not considered acceptable)
* Female participants not of child-bearing potential (that is, are postmenopausal or permanently sterilized [such as, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy]). Such participants will not be required to use contraception but must test negative for pregnancy at the time of enrollment
* Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) or spontaneous amenorrhea for 6 to 12 months, with follicle stimulating hormone (FSH) ≥40 milli-international units per milliliters (mIU/mL)
* Female participants who have undergone sterilization by tubal ligation agree to use a condom in conjunction with spermicidal gel, foam, cream, film or suppository from the time of screening until 3 months after the last dose of investigational product. Such participants must also test negative for pregnancy at the time of enrollment
* Have a body mass index (BMI) of 18.5 to 32.0 kilograms per meters squared (kg/m^2), inclusive, at screening
* Have clinical laboratory test results within the normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures and are willing to follow study restrictions
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are currently enrolled in or have completed or discontinued within the last 30 days from a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to Glucagon-like peptide 1 (GLP-1) -related compounds including dulaglutide, or any components of the formulation
* Are persons who have previously completed or withdrawn from this study or any other study investigating dulaglutide in the 3 months prior to screening or have received glucagon-like peptides or incretin mimetics in the 3 months prior to screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure (after at least 5 minutes sitting) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder, for example relevant esophageal reflux or gall bladder disease, or any gastrointestinal disease which impacts gastric emptying (such as, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by GLP-1 analogs. Participants with dyslipidemia, and participants who had cholecystolithiasis (removal of gall stones) and/or cholecystectomy (removal of gall bladder) in the past, with no further sequelae, may be included in the study at the discretion of the screening physician
* Show evidence of significant active neuropsychiatric disease
* Have family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Have used or intend to use over-the-counter medication other than acetaminophen within 7 days prior to dosing or prescription medication (with the exception of vitamin/mineral supplements and/or hormone replacement therapy [HRT]) within 14 days prior to dosing
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females), or are unwilling to adhere to the alcohol restrictions (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Smoke more than 10 cigarettes (or equivalent in nicotine) per day, and are unwilling to refrain from smoking on the day of dulaglutide administration or are unable to abide by clinical research unit (CRU) restrictions
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Syringe First, Then Auto-injector: First Intervention:
  Dulaglutide: A single dose of 1.5 milligrams (mg) dulaglutide administered subcutaneously (SC) by manual syringe.
  There was a washout period of at least 28 days between treatment periods.
  Second intervention:
  Dulaglutide: A single dose of 1.5 mg dulaglutide administered SC by auto-injector.
- Auto-injector First, Then Manual Syringe: First Intervention:
  Dulaglutide: A single dose of 1.5 milligrams (mg) dulaglutide administered subcutaneously (SC) by auto-injector.
  There was a washout period of at least 28 days between treatment periods.
  Second intervention:
  Dulaglutide: A single dose of 1.5 mg dulaglutide administered SC by manual syringe.
Period: First Intervention
Arm/Group | Manual Syringe First, Then Auto-injector | Auto-injector First, Then Manual Syringe
Started | 26 | 24
Received at Least 1 Dose of Study Drug | 26 | 24
Completed | 23 | 23
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Period: Washout Period of at Least 28 Days
Arm/Group | Manual Syringe First, Then Auto-injector | Auto-injector First, Then Manual Syringe
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Manual Syringe First, Then Auto-injector | Auto-injector First, Then Manual Syringe
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of dulaglutide.
Groups:
- Entire Study Population: All participants who received at least one 1.5-milligram (mg) dose of dulaglutide administered subcutaneously via manual syringe or auto-injector.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 35
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC[0-336]) for Dulaglutide
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least 1 dose of dulaglutide and have evaluable dulaglutide concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hours per milliliters
Groups:
- Auto-injector: Dulaglutide: Single dose of 1.5 milligrams (mg) dulaglutide administered subcutaneously (SC) by auto-injector in one of two study periods separated by a minimum 28 day washout period.
- Manual Syringe: Dulaglutide: Single dose of 1.5 milligrams (mg) dulaglutide administered subcutaneously (SC) by manual syringe in one of two study periods separated by a 28 day minimum washout period.
Arm/Group | Auto-injector | Manual Syringe
Number analyzed (Participants) | 47 | 47
nanograms times hours per milliliters | 14700 (22) | 14300 (24)

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) for Dulaglutide
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least 1 dose of dulaglutide and have evaluable dulaglutide concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Auto-injector | Manual Syringe
Number analyzed (Participants) | 47 | 48
nanograms per milliliter (ng/mL) | 91.1 (31) | 88.2 (32)

3. Secondary Outcome: Pharmacokinetics: Time to Maximum Concentration (Tmax) for Dulaglutide
Time Frame: Predose to 336 hours postdose
Population: Participants who received at least 1 dose of dulaglutide with evaluable concentration-time data.
Measure: Median (Full Range); unit: hours
Arm/Group | Auto-injector | Manual Syringe
Number analyzed (Participants) | 47 | 48
hours | 48.0 [24.0 to 96.0] | 48.0 [24.0 to 96.0]

ADVERSE EVENTS:
Arm/Group | Auto-injector | Manual Syringe
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/49
Other Adverse Events (participants affected / at risk) | 18/47 | 18/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-injector (N=47) | Manual Syringe (N=49)
Constipation (Gastrointestinal disorders) | 5 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (4)
Asthenia (General disorders) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 8 (8)
Headache (Nervous system disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days